CLINICAL TRIAL: NCT06668259
Title: Intensive Longitudinal Assessment of Stress and Stress-related Concepts Across a Behavioral Weight Loss Intervention: INSTANT Study
Brief Title: Intensive Longitudinal Assessment of Stress and Stress-related Concepts Across a Behavioral Weight Loss Intervention
Acronym: INSTANT
Status: Recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Chelsea L. Kracht, PhD, Assistant Professor, University of Kansas Medical Center
Other Study IDs: STUDY00160436; 5P20GM144269-03 (NIH)
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Individual Stress and Weight Loss
Keywords: stress; weight loss; EMA; weight gain; cortisol; surveys
MeSH Terms: conditions — Weight Loss; Weight Gain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Salivary cortisol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Examine the association between variability in individual stress and related concepts with weight loss, physical activity, and sleep across a behavioral weight loss program

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in a community-based weight loss program centered in a metropolitan area of a Midwest state. Based on this criteria, we will anticipate participants are greater than 18 years of age, and have obesity.
* Must own a smart phone and be willing to download the mobile application to receive text messages

Exclusion Criteria:

* Report a current medical condition or treatment for a medical condition that could affect body weight.
* Current psychological condition (including clinically diagnosed depression) that is untreated, hospitalization for a psychological condition within the past 12 months, or not being on a stable dose of treatment for at least 6 months.
* Is not fluent in writing or speaking the English language.
* Mobility limitations so they are unable to perform physical activity.
* Family member currently enrolled in the study or has a family member that previously participated in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who are enrolled in a community-based weight loss program centered in a metropolitan area of a Midwest state will be eligible to participate
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Weight (kg) | 0 Weeks, 6 Weeks, 12 Weeks, and 26 Weeks
  Weight will be measured using a digital scale in kg to the nearest 0.1 kg.
Physical Activity | 0 Weeks, 6 Weeks, 12 Weeks, and 26 Weeks
  Physical activity will be device-measured using an ActiGraph accelerometer. Participants will wear the accelerometer on their wrist for 14 consecutive days. Accelerometer will only be removed for water-based activities.
Sleep | 0 Weeks, 6 Weeks, 12 Weeks, and 26 Weeks
  Sleep will be device-measured using an ActiGraph accelerometer. Participants will wear the accelerometer on their wrist for 14 consecutive nights.
Stress-related Concepts (EMA) | 0 Weeks, 6 Weeks, 12 Weeks, and 26 Weeks
  Stress-related concepts are measured by surveys of daily coping ability, stress, and affect assessed by Ecological Momentary Assessments (EMA). For daily coping, participants will be asked about their ability to cope with stress, on a scale from 0-10 with 10 indicating completely able to cope. For stress participants will be asked about their current stress level, on a scale from 0-10 with 10 indicating the highest stress. Affect will be assessed through 5 questions related to their current feeling of happiness, frustration, stress, anger, sadness, and calm/relaxed.

SECONDARY OUTCOMES:
Cortisol (mg/mL) | 0 Weeks, 6 Weeks, 12 Weeks, and 26 Weeks
  Collected via salivary collection methods

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Fairway North, Fairway, Kansas
  - Kirmayer Fitness Center, Kansas City, Kansas

IPD SHARING:
Plan to Share IPD: Yes
Clinical data will be shared with controlled access in NIDDK Central Repository for general research use
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 1 year after publication with no end date.
Access Criteria: Data will be stored in the NIDDK Central Repository data repository. Other requests for data and further information can be made to the PI, who will follow appropriate channels to distribute the data.